CLINICAL TRIAL: NCT04860674
Title: A Prospective, Single-arm, Phase II Study of PD-1 Inhibitor Combined With Ifosfamide, Carboplatin, and Etoposide (ICE) in the Treatment of Relapsed/Refractory Gray Area Lymphoma
Brief Title: A Prospective Study of PD-1 Inhibitor Combined With ICE in the Treatment of Relapsed/Refractory Gray Area Lymphoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Principal Investigator, Yang haiyan, Director, Zhejiang Cancer Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PICE
Record Dates: First submitted 2021-02-02; First posted 2021-04-27 (Actual); Last update posted 2021-04-27 (Actual); Status verified 2021-04

CONDITIONS: Gray Zone Lymphoma; Relapse/Recurrence; Chemotherapy Effect
MeSH Terms: conditions — Recurrence | interventions — Carboplatin; Etoposide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PD-1+ICE (Experimental): PD-1 inhibitor combined with icyclophosphamide, carboplatin, etoposide chemotherapy
  Interventions: Drug: PD-1 inhibitor +ICE

INTERVENTIONS:
Drug: PD-1 inhibitor +ICE — PD-1 inhibitor (tirelizumab) combined with ifosfamide, carboplatin and etoposide (ICE) regimen
  Other Names: Icyclophosphamide; carboplatin; etoposide

SUMMARY:
There are no standard chemotherapy regimens for relapse/refractory gray area lymphoma. The programmed cell death ligand 1 (PD-L1) encoding gene is located in 9p24.1, so it is speculated that the programmed cell death pathway plays an important role in gray area lymphoma formation by evading immune surveillance in GZL.The purpose of this study was to evaluate the efficacy and safety of PD-1 monoclonal antibody combined with ICE in the treatment of patients with relapsed/refractory gray area lymphoma.

DETAILED DESCRIPTION:
The purpose of this study was to evaluate the efficacy and safety of PD-1 monoclonal antibody combined with ICE in the treatment of patients with relapsed/refractory gray zone lymphoma. The main study endpoint is the Objective Response Rate (ORR), including Complete Remission Rate (CRR) and Partial Remission Rate (PRR), was evaluated according to Lugano2014 lymphoma efficacy evaluation criteria.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary participation in the clinical study: fully understand and know the study and sign the informed consent form in person;Willing to follow and able to complete all testing procedures.
2. Age: 18~70 years old (inclusive), both male and female.
3. Histopathologically confirmed gray zone lymphoma (between HD and DLBCL).
4. Recurrent or refractory disease after receiving at least first-line standard chemotherapy (refractory is defined as chemotherapy not reaching CR or PR).
5. ECOG score is 0-2 points.
6. Expected survival of at least 3 months.
7. There must be at least one evaluable or measurable lesion that meets the Lugano2014 criteria.
8. Sufficient organ and bone marrow function, no serious hematopoietic dysfunction, abnormal heart, lung, liver, kidney function and immune deficiency
9. Left ventricular ejection fraction (LVEF) ≥ 50% in cardiac function examination.
10. Serum pregnancy test was negative and effective contraceptive measures were taken from the signing of informed consent until 6 months after the use of the last chemotherapy.
11. Thyrotropin (TSH) or free thyroxine (FT4) or free triiodothyronine (FT3) were within the range of ±10% of normal values.
12. There was no evidence that subjects had difficulty breathing at rest and their pulse oximetry at rest was >95%.
13. Subjects must confirm the first forced expiratory volume (FEV1)/forced expiratory volume (FVC) >60% by pulmonary function test, unless large mediastinal mass compression fails to meet this standard;Carbon monoxide dispersion (DLCO), FEV1 and FVC all exceeded the predicted value by more than 50%.
14. Subjects who had received previous anti-tumor therapy were admitted only after the toxicity of previous therapy returned to CTCAE V5.0 level ≤1 or baseline;Class 2 toxicity (such as neurotoxicity, alopecia, and hearing loss) that was irreversible and not expected to worsen during the study period due to prior antitumor therapy were assessed by the investigator and were eligible for inclusion.

    -

Exclusion Criteria:

1. Central nervous system involvement.
2. Participating in other clinical studies, or administering the first study drug less than 4 weeks after the end of treatment in the previous clinical study.
3. Had other malignant tumors in the past 5 years, except basal cell carcinoma of the skin, squamous cell carcinoma of the skin, carcinoma in situ of the breast, and carcinoma in situ of the cervix after radical treatment.
4. The last antitumor treatment was less than 3 weeks after the first administration of the drug in this study, including chemotherapy, immunotherapy, radiotherapy, and biotherapy (tumor vaccines, cytokines, or growth factors for cancer control).
5. Previous allogeneic hematopoietic stem cell transplantation or prior ASCT or CAR-T therapy within 1 month prior to initial dosing of the investigational drug.
6. Have previously received PD-1 or PD-L1 targeted therapy.
7. A history of severe hypersensitivity to monoclonal antibodies.
8. Major surgery was performed within 28 days prior to the start of study treatment.
9. In this study, the patients received anti-tumor Chinese herbal medicine or proprietary Chinese medicine within 7 days before the first medication.
10. Live vaccine (except attenuated influenza vaccine) was administered within 28 days before the first administration.
11. Patients with a known history of Human Immunodeficiency Virus (HIV) infection and/or acquired Immunodeficiency syndrome.
12. Patients with active history of autoimmune disease or blood body autoimmune disease and patients with high risk of recurrence, including but not limited to the immune related neuropathy, multiple sclerosis, autoimmune, demyelinating neuropathy, GBS, myasthenia gravis, systemic lupus erythematosus (sle), scleroderma, connective tissue disease, inflammatory bowel cancer (including crohn's disease and ulcerative colitis), autoimmune hepatitis, toxic epidermal necrosis release or Stevens Johnson syndrome.
13. Corticosteroid (prednisone >10mg/d or equivalent) or other immunosuppressive systemic therapy should be used within 14 days prior to the first administration of the study drug.
14. Patients with active chronic hepatitis B or active hepatitis C.
15. Have active tuberculosis.
16. Present with interstitial pulmonary disease or non-infectious pneumonia.
17. Active infections requiring systematic anti-infective treatment, including but not limited to bacterial, fungal or viral infections.
18. Pregnant or lactating women.
19. Patients with New York Heart Association (NYHA) grade III or IV heart failure, unstable angina, severe poorly controlled ventricular arrhythmias, and electrocardiographic findings of acute ischemia or myocardial infarction during the preceding 6 months were screened.
20. QTCF interphase >480 Msec, unless secondary to bundle branch block.
21. Have an uncontrollable combined disease, including but not limited to uncontrollable hypertension, active peptic ulcer or hemorrhagic disease.
22. People with previous psychiatric history;Having no capacity or limited capacity.
23. The underlying condition of the patient, as determined by the investigator, may increase the risk of receiving the study drug, or may cause confusion about the perceived toxicity and its assessment.
24. Patients considered by other investigators to be unsuitable for this study. -

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-05-01 (Estimated); Primary Completion 2024-04-01 (Estimated); Study Completion 2024-04-01 (Estimated)

PRIMARY OUTCOMES:
ORR | From enrollment until date of completion of chemotherapy, at the end of cycle 6 (each cycle is 21 days)
  overall response rate

SECONDARY OUTCOMES:
PFS | From date of first day of treatment until the date of first documented progression, assessed up to 24 months
  Progression Free Survival
OS | From date of first day of treatment until the date of first documented date of death from any cause, assessed up to 24 months
  Overall Survival
AE and SAE | From data of first day of treatment until 30 day after last treatment
  Adverse event and serious adverse event

CONTACTS AND LOCATIONS:
Overall Officials: Cong Li, Principal Investigator — Zhejiang Cancer Hospital

IPD SHARING:
Plan to Share IPD: No
The IPD is related to participants' privacy